CLINICAL TRIAL: NCT07389902
Title: The Impact of Conversational Approaches in Pediatric Robot-Mediated Interventions on Children's Responses in Hospital Settings: A Comparative Study of Rule-Based vs. LLM-Based Systems
Brief Title: Impact of Conversational Approaches in Pediatric Social Robot-Mediated Interventions
Acronym: PRIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMC 2025-09-101-003
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Patients; Pediatric Patients in Hospital Settings; Hospitalized Children
Keywords: Child-robot interaction; Social robot; Pediatric hospitalization; Large language models; Human-robot interaction; Pediatric care

STUDY DESIGN:
Intervention Model Description: Between-subjects factor: Robot dialogue type Within-subjects factor: Content type
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rule-Based Robot Dialogue (Experimental): Participants interact with LIKU robot using pre-programmed, rule-based dialogue responses. Each participant completes two activity sessions (emotional support content and safety education content) in randomized order.
  Interventions: Behavioral: Robot-Mediated Emotional Support Activity; Behavioral: Robot-Mediated Safety Education Activity
- LLM-Based Robot Dialogue (Experimental): Participants interact with LIKU robot using large language model-generated dialogue responses. Each participant completes two activity sessions (emotional support content and safety education content) in randomized order.
  Interventions: Behavioral: Robot-Mediated Emotional Support Activity; Behavioral: Robot-Mediated Safety Education Activity

INTERVENTIONS:
Behavioral: Robot-Mediated Emotional Support Activity — 10-15 minute structured activity focusing on emotional recognition, expression, and regulation through storytelling, discussion, and artistic activities (drawing, physical expression) with the LIKU social robot
Behavioral: Robot-Mediated Safety Education Activity — 10-15 minute structured activity focusing on safety awareness and emergency response behaviors through educational videos, discussions, and hands-on activities (crafts, physical practice) with the LIKU social robot

SUMMARY:
This study examines how different robot dialogue systems (rule-based vs. large language model-based) and content types (emotional support vs. safety education) affect pediatric patients' responses during hospital-based robot-mediated interventions.

Approximately 60 pediatric patients aged 2-9 years will be randomly assigned to interact with a social robot (LIKU) using either rule-based or LLM-based dialogue. Each child will participate in two activity sessions (emotional content and safety content) in randomized order.

Primary outcomes include child engagement, emotional responses, robot perception, and activity preferences, assessed through standardized questionnaires (UEQ, Godspeed), child interviews, and behavioral observations. Additionally, 5 experts will evaluate content appropriateness and safety.

This pilot study aims to provide foundational data for developing personalized pediatric robot programs in hospital settings, optimizing both dialogue approaches and content design based on individual child characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 2-9 years
* Currently admitted to or visiting Samsung Medical Center pediatric ward or outpatient clinic
* Capable of cognitive communication as determined by experienced medical staff
* Written informed consent from parent/legal guardian obtained
* Verbal assent from child obtained (developmentally appropriate)
* Not in acute emergency situation
* Able to engage in stable interaction for at least 5 minutes in hospital environment

Exclusion Criteria:

* Diagnosis of moderate to severe developmental delay (language or cognitive) documented in medical records
* Currently in isolation treatment (e.g., due to infectious disease)
* Experiencing acute pain, fever, or medical procedures that make study participation difficult
* Parent/guardian or child declined participation or withdrew consent

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Child Engagement Level | Immediately following each intervention session (assessed within 1 hour post-session)
  Behavioral observation checklist assessing attention to robot, participation in activities, and task involvement. Scored by trained observers using standardized coding scheme based on video recordings.
User Experience | Immediately following each intervention session (approximately 5 minutes post-session)
  User Experience Questionnaire (UEQ) - standardized 7-point semantic differential scale measuring six dimensions: attractiveness, perspicuity, efficiency, dependability, stimulation, and novelty of robot interaction.
Robot Perception | Immediately following each intervention session (approximately 5 minutes post-session)
  Godspeed Questionnaire Series - standardized scale measuring five dimensions of robot perception: anthropomorphism, animacy, likeability, perceived intelligence, and perceived safety.

SECONDARY OUTCOMES:
Content Appropriateness | Within 2 weeks of session completion via video review
  Expert evaluation using 5-point Likert scale assessing developmental appropriateness, educational fit, robot speech pacing, content clarity, and activity flow. Evaluated by 5 pediatric development experts through video review.
Activity Preference | Immediately following completion of both intervention sessions (approximately 5 minutes)
  Child interview using picture cards to identify preferred activities and content types (emotional support vs safety education). Children select and explain their preferences.
Content Comprehension | Immediately following each intervention session (approximately 3 minutes)
  Child interview assessing understanding of activity content, key messages, and learning points from each session using age-appropriate questions.
Robot Relationship Quality | Immediately following intervention sessions (approximately 5 minutes)
  Child interview and behavioral observation assessing perceived intimacy with robot, emotional attachment, social bonding, and willingness to interact with robot again.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No